CLINICAL TRIAL: NCT03258268
Title: A 26-week, Multicenter, Controlled Trial of the Glycemic Outcomes of Individualized Treatment Support in Patients With Type 2 Diabetes
Brief Title: Easy Diabetes Treatment Study 1
Acronym: EASY-1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Läkarexpressen AB (Industry)
Collaborators: Region Skane (Other); Lund University (Other); Region Halland (Other); Västra Götalandsregionen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EASY-1
Record Dates: First submitted 2017-08-20; First posted 2017-08-23 (Actual); Last update posted 2020-10-05 (Actual); Status verified 2020-09

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Multicenter, randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: A double-blind design is not feasible due to the need for physicians to use respectively not use the EASY DSS.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care with DSS (Experimental): Patients will receive standard of care with a board certified physician with EASY DSS.
  The choice of treatment will be made by the investigator. In the investigational arm this will be based on the clinical judgment of the investigator supplemented with support from the EASY DSS and in the control arm this will be based on the clinical judgment of the investigator alone.
  Interventions: Device: Standard of Care with EASY DSS
- Standard of Care without DSS (Active Comparator): Patients will receive standard of care with a board certified physician without EASY DSS.
  The choice of treatment will be made by the investigator. In the investigational arm this will be based on the clinical judgment of the investigator supplemented with support from the EASY DSS and in the control arm this will be based on the clinical judgment of the investigator alone.
  Interventions: Other: Standard of Care without EASY DSS

INTERVENTIONS:
Device: Standard of Care with EASY DSS — The EASY DSS is a software tool designed to process and analyze data to facilitate individualized treatment suggestions for type 2 diabetes patients.
  Patients will receive standard of care with a board certified physician with EASY DSS.
  The choice of treatment will be made by the investigator. In the investigational arm this will be based on the clinical judgment of the investigator supplemented with support from the EASY DSS and in the control arm this will be based on the clinical judgment of the investigator alone.
  Arms: Standard of Care with DSS
Other: Standard of Care without EASY DSS — Patients will receive standard of care with a board certified physician without EASY DSS.
  The choice of treatment will be made by the investigator. In the investigational arm this will be based on the clinical judgment of the investigator supplemented with support from the EASY DSS and in the control arm this will be based on the clinical judgment of the investigator alone.
  Arms: Standard of Care without DSS

SUMMARY:
A 26-week, multicenter, parallel two-arm, randomized controlled trial of the glycemic outcomes of individualized treatment support in patients with type 2 diabetes. The primary objective of the trial is to confirm the superiority of standard of care with EASY DSS versus standard of care without EASY DSS in terms of glycemic control in patients with type 2 diabetes with ongoing treatment with any antidiabetic drug(s).

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained before any trial-related activities. Trial-related activities are any procedures that are carried out as part of the trial, including activities to determine suitability for the trial
* ≥ 18 years of age at the time of signing informed consent
* Type 2 diabetes (diagnosed clinically) ≥ 6 months prior to screening
* HbA1c ≥ 7.0 [58 mmol/mol] by central laboratory analysis
* Stable daily treatment with any single antidiabetic drug or any combination of antidiabetic drugs for at least 90 days prior to screening (dose adjustment ±10% of insulin dose and temporary dose correction because of e.g. infection are allowed)

Exclusion Criteria:

* Previous participation in this trial. Participation is defined as informed consent.
* Currently participating in other clinical trials for diabetes
* Type 1 diabetes diagnosed clinically and/or by the presence of diabetes-associated autoantibodies
* History of diabetic ketoacidosis or hyperosmolar hyperglycemic state
* Corticosteroid-induced or pancreatitis-induced diabetes
* History of chronic or acute pancreatitis
* Known or suspected substance abuse
* Pregnancy
* Anticipated change in concomitant medication, which, in the opinion of the investigator, could interfere with the glucose metabolism (e.g. systemic corticosteroids or statins)
* Uncontrolled hypertension (systolic blood pressure > 180 mmHg and/or diastolic blood pressure > 100 mmHg)
* Renal failure stage 5, defined as (estimated or exact) glomerular filtration rate < 15 mL/min/1.73m2
* Recent or planned major surgery (such as gastric bypass operation)
* Major psychiatric disorders, mental incapacity, unwillingness or language barrier precluding adequate understanding of the trial procedure or cooperation with the trial site personnel
* Life-threatening disease including malignant neoplasms and medical history of malignant neoplasms within the last 5 years (except basal and squamous cell skin cancer)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 311 (Actual)
Dates: Start 2017-08-07 (Actual); Primary Completion 2019-12-12 (Actual); Study Completion 2019-12-19 (Actual)

PRIMARY OUTCOMES:
HbA1c | 26 weeks
  Change from baseline HbA1c

SECONDARY OUTCOMES:
Fasting plasma glucose | 26 weeks
  Change from baseline in fasting plasma glucose (FPG)
Achieving treatment target | 26 weeks
  Meeting treatment target of HbA1c < 7% (53 mmol/mol)
Hypoglycemia | 26 weeks
  Meeting treatment target of HbA1c < 7% (53 mmol/mol) without severe or clinically significant hypoglycemic episodes

CONTACTS AND LOCATIONS:
Overall Officials: Damon Tojjar, MD, Principal Investigator — Lund University
Locations (3):
- Sweden (3):
  - Region Halland, Hålland
  - Region Skåne, Skåne
  - Västra Götalandsregionen, Västra Götaland

IPD SHARING:
Plan to Share IPD: No